CLINICAL TRIAL: NCT00766038
Title: A Phase II, Randomized Controlled Trial of Recombinant Human Growth Hormone During Rehabilitation From Traumatic Brain Injury.
Brief Title: Recombinant Human Growth Hormone During Rehabilitation From Traumatic Brain Injury.
Acronym: Growth-TBI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Baylor Health Care System (Other)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Professor of Neurology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTTBIMS-GH RCT; NIDRR H133A07002708; Pfizer GA62816O
Record Dates: First submitted 2008-09-30; First posted 2008-10-03 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Traumatic Brain Injury
Keywords: Mood disorders; Cognitive disorders; Fatigue; Metabolic disorders
MeSH Terms: conditions — Brain Injuries, Traumatic; Mood Disorders; Cognitive Dysfunction; Fatigue; Metabolic Diseases | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The GH treatment arm will receive a starting dose of 400 microgramsg/day, with increases (or decreases) in dose by 100-200 micrograms/day each month, monitoring for side effects, until goal IGF-1 (in the upper quartile of the range for age and body weight) is reached up to maximum dose of 1,000 microgramsg/day. Dose adjustments may be modified by the investigators for participants receiving oral estrogens or other circumstances know to influence GH dosing or atypical responses to treatment.
  Interventions: Drug: Recombinant human Growth Hormone
- 2 (Placebo Comparator): Doses for participants receiving placebo will also be adjusted monthly to maintain the blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant human Growth Hormone — 400 micrograms/day SC for 6 months. Dose adjusted based on serum IGF-1 measurements
  Other Names: Somatotropin; Genotropin(R); HGH
  Arms: 1
Drug: Placebo — SC injection daily
  Arms: 2

SUMMARY:
Growth Hormone (GH) deficiency, defined by insufficient GH response to a variety of stimulating compounds, is found in 20-35% of adults who suffer traumatic brain injuries (TBI) requiring inpatient rehabilitation1. However, there is no accepted gold standard for diagnosing GH deficiency in this population. Further, the major effector molecule of the somatotropic axis, Insulin-Like Growth Factor-1 (IGF-1) has recently been recognized as an important neurotrophic agent. Since most repair and regeneration after TBI occurs within the first few months after injury, absolute or relative deficiencies of GH and IGF-1 in the subacute period after TBI are potentially important factors why some patients fail to make a good functional recovery. The proposed study is a randomized, double-blind, placebo-controlled trial of rhGH, starting at 1 month post TBI, continuing for 6 months.

This study has one primary hypothesis, that treatment with recombinant human Growth Hormone (rhGH) in the subacute period after TBI results in improved functional outcome 6 months after injury. As secondary hypotheses, we will investigate what is the optimal method to diagnose GH deficiency in TBI survivors and study the relationship between GH deficiency and insufficiency and functional recovery.

DETAILED DESCRIPTION:
1. Patient selection and enrollment. Participants will be recruited into the study from subjects admitted for acute inpatient rehabilitation in the North Texas Traumatic Brain Injury Model Systems (NT-TBIMS) affiliated rehabilitation units. Our goal is to enroll participants who have the potential for neuroregeneration, but who suffered a sufficiently severe injury that the chance of full recovery (to normal pre-injury function) is low. Over a 4 year enrollment period, we plan to randomize 168 subjects into the study (with the anticipation that 71 will complete each arm of the trial).

Inclusion Criteria

1. Non-penetrating TBI
2. Age 18 - 50 years.
3. Admission to a North Texas Traumatic Brain Injury Model System-affiliated rehabilitation unit within 8 weeks of injury. Enrollment in TBI-MS database not required.
4. Randomization within 2 - 10 weeks of injury.
5. Rancho Los Amigos Rating IV or better at the time of randomization. Should not be at Rancho IV level for more than 4 weeks before randomization.

5. GH deficiency diagnosed by either of the following two criteria:

1. . Peak GH response to L-arginine stimulation test < 1.4 microg/L; or
2. . Plasma IGF-1 level 1 SD below the expected median for age and body weight. 6. Availability of caregiver to oversee administration of medications. 7. Reasonable expectation for completion of outcome measures 8. Residence inside the United States.

Exclusion Criteria:

1. History of pre-existing neurologic disease (such as epilepsy, brain tumors, meningitis, cerebral palsy, encephalitis, brain abscesses, vascular malformations, cerebrovascular disease, Alzheimer's disease, multiple sclerosis, or HIV-encephalitis)
2. History of premorbid disabling condition that interfere with outcome assessments
3. Contraindication to rhGH therapy. (hypersensitivity to rhGH or any of the components of the supplied product, including metacresol, glycerin, or benzyl alcohol)
4. Penetrating traumatic brain injury
5. Diabetes mellitus.
6. Obesity (BMI > 30).
7. Active infection.
8. Active malignant disease.
9. Acute critical illness, heart failure, or acute respiratory failure
10. Previous hospitalization for TBI > 1 day
11. Membership in a vulnerable population (prisoner)
12. Pregnancy. Women of childbearing age will be given a pregnancy test during screening to exclude pregnancy.
13. Lactating females

We will measure baseline IGF-1 as well as carry out L-arginine GH stimulation tests prior to entry into the study, and measure IGF-1 levels again at completion of the treatment phase.

2. Treatment. After obtaining informed consent, we will measure IGF-1 levels as well as perform dynamic GH testing. Eligible patients will be randomization in a double-blind fashion to (Group 1) rhGH subcutaneously or (Group 2) placebo. The GH treatment arm will receive a starting dose of 400 microg/day, with increases (or decreases) in dose by 100-200 microg/day each month, monitoring for side effects, until goal IGF-1 (in the upper quartile of the range for age and body weight) is reached up to maximum dose of 1,000 microg/day. Dose adjustments may be modified by the investigators for participants receiving oral estrogens or other circumstances know to influence GH dosing or atypical responses to treatment. Doses for participants receiving placebo will also be adjusted monthly to maintain the blinding.

The treatment will be overseen by a board certified endocrinologist (Dr. Auchus), according to practice guidelines recently released by the Endocrine Society "Clinical Guidelines for Evaluation and Treatment of Adult Growth Hormone Deficiency". The principle is that therapy is started at a relatively low dose and increased monthly, adjusting for the occurrence of adverse effects. In this study, to accommodate both GH-deficient and GH-sufficient strata, the treatment goal is serum IGF-1 as close as possible to the upper limit for the age-adjusted reference range without exceeding this normal range.

The objective of randomization is to produce study groups comparable with respect to known and unknown risk factors, to remove investigator bias in the recruitment and allocation of participants and to guarantee that statistical tests have valid significance levels. To balance factors that may influence treatment outcome, randomization will be stratified and blocked, by two factors:

1. Age (< 35 years vs. > 35 years)
2. Severity of injury (duration of post-traumatic amnesia < 20 days vs. > 20 days).

   Each combination of factors forms a stratum and randomization is allocated within each stratum.

   GH Stimulation Test: After obtaining informed consent, an 18 - 20 g IV catheter is placed in a forearm vein. 5 ml of blood is sampled at baseline, and afterwards L-arginine is infused over 30 minutes (in 100 mL NS, dose 0.5 g/kg up to a maximum of 30 g). Blood is sampled at 30, 60, and 90 minutes after starting the infusion of the L-arginine. All blood samples are centrifuged and serum frozen at -20oC within 15 minutes of collection. All serum specimens are assayed for glucose and GH. Growth Hormone deficiency is defined as a peak response to arginine infusion < 1.4 ng/mL. Growth Hormone insufficiency is defined as peak GH response < For IGF-1 levels, we will use the age and gender normative data based on 3,961 healthy subjects.
3. Safety Assessments. Safety will be assessed by clinical evaluations at 1, 2, 3, and 4.5 months after initiating therapy. At these evaluations participants and their caregivers will be asked about possible adverse effects of GH treatment, including fluid retention, paresthesias, joint stiffness, peripheral edema, arthralgias, and myalgias. Additionally, blood will be obtained for assessment of glucose, free T4, lipid profile, and insulin level. The dose of GH (or placebo) will be adjusted by the study physician depending on the occurrence and severity of adverse effects.
4. Outcome Measures. Table 3 summarizes the functional and neuropsychologic tests we will use to assess outcome in our study. This battery of measures was developed by the NCMRR TBI Clinical Trials Network to maximize power in TBI clinical trials compared to a single measure alone. These measures are designed to capture a broad perspective of functional and cognitive parameters that are important following TBI, and utilizes scales that have a long history in TBI research. Further, there is convincing evidence that they can be reliably administered 6 - 12 month after injury.
5. Biochemical tests. Plasma GH and IGF-1 levels will be measured by the Clinical Contracts Research Laboratories at UT Southwestern Medical Center (CLIA ID No. 45D0659587), using commercially-available immunoassays. This laboratory will also carry out the safety lab assessments (glucose, insulin, free T4, lipid profile. Results will be available within 1 week to allow randomization within the time window, and to allow dose adjustments in a timely fashion.
6. Statistical Analysis and Sample size calculation. This is a Phase II study, designed to assess feasibility and obtain information about dosing efficacy and magnitude of effect. There are two features of the study design that are relatively novel to TBI clinical trials, which merit some introduction. The first is the use of a futility (non-inferiority) design, and the second is the use of a composite outcome statistic.

The goal of Phase II studies is to provide information about side effects and toxicities in the type of patients for whom the treatment is intended, determine the logistics of administration, provide estimates of treatment costs, and obtain some information about expected effect size. For reasons discussed above, we believe that such information is not yet available regarding the use rhGH in the early phase after TBI, and that a Phase II study designed to obtain this information is warranted. Drugs that remain promising after Phase II studies generally proceed to Phase III clinical trials, which typically require many hundreds of patients and are usually conducted at multiple centers and at great expense.

Futility design trials were pioneered in cancer chemotherapy studies, and have recently been used in Phase II clinical trials of neurological disorders such as Parkinson's disease and stroke. A traditionally designed study focuses on efficacy, with a null hypothesis that the treatment arms are equivalent. In such studies, the assumption is that a false positive result is riskier than a false negative result (that it is riskier to falsely assume than an ineffective therapy works than it is to discard a potentially effective treatment). In such studies, it is customary to set alpha at 0.05 (the likelihood of a false positive result less than 5%), and beta at 0.2 (the likelihood of a false negative result--that a beneficial effect will be missed is less than 20%). A futility design incorporates the view that in the early phases of clinical development of a new therapy, it is in fact riskier to discard a potentially useful treatment than it is to fail to definitively identify efficacy, since that can only be done in a phase III study. Thus, in a phase II futility study the null hypothesis is that treatment has promise and will therefore produce results exceeding a meaningful threshold. Thus, alpha of 0.1 (as set in our study) in a futility study means that the chance of beneficial effect being missed is less than 10%. In a futility design, if the efficacy threshold is not met, the null hypothesis is rejected and further study of the treatment is considered futile42. Thus, for the primary hypothesis, the design of our study is that of a futility (non-superiority) study, powered to not reject a potentially useful therapy, rather than prove efficacy.

The second relatively novel feature of our study is the use of a composite outcome statistic. A composite outcome statistic takes into account the fact that in a complex disorder such as TBI, there are multiple domains of dysfunction, and a single scale (such as the GOS-E or a given neuropsychometric test) may not be optimally sensitive to identify functionally important deficits in all patients. There are several mathematical approaches to the need to compare two groups with respect to more than one outcome. The options available include using Bonferroni or other adjustments for multiple comparisons, reducing the dimensions of the problem by averaging the outcomes, or applying a global test based on a multiple correlated binary outcomes43,44. Of these, the latter approach has been found to be useful in a variety of clinical settings. Incorporating several different measures, which although correlated measure different domains of dysfunction after TBI, significantly lowers the sample size required. We have elected to use a composite outcome statistic developed by the NIH TBI Clinical Trials Network, which will be used in the Citocholine Brain Injury Treatment (COBRIT) study. This measure was developed by a subcommittee of the NIH network that included clinicians, neuropsychologists, and biostatisticians, including Dr. Diaz-Arrastia and Dr. Sureyya Dikmen (who will serve in the DSMB for this trial). In our study, the use of a composite statistic lowers the sample size from 228 to 164.

All participants in the GH treatment arm may not achieve goal serum IGF-1 values in the first month, yet data will be analyzed in an intention-to-treat manner.

Primary Hypothesis:

1. . Treatment with recombinant human Growth Hormone (rhGH) in the subacute period after TBI results in improved functional outcome 6 months after injury, as measured by the Composite Outcome Score of the TBI Clinical Trials Network .

   Secondary Hypotheses:
2. . Treatment with rhGH results in increased IGF-1 levels.
3. . rhGH treatment results in improved bone mineral density and lean body mass 6 months after injury.
4. . Benefits of rhGH treatment persist up to 1 year after injury
5. . Low GH response to L-arginine stimulation at baseline is associated with poor functional outcome.
6. . Low IGF-1 levels at baseline are associated with poor functional outcomes.
7. . rhGH treatment is more effective in patients who have low IGF-1 levels at baseline.
8. . rhGH treatment is more effective in patients who have low GH response to L-Arginine stimulation at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Non-penetrating TBI
2. Age 18 - 50 years.
3. Admission to a North Texas Traumatic Brain Injury Model System-affiliated rehabilitation unit within 8 weeks of injury. Enrollment in TBI-MS database not required.
4. Randomization within 2 - 10 weeks of injury.
5. Rancho Los Amigos Rating IV or better at the time of randomization. Should not be at Rancho IV level for more than 4 weeks before randomization.
6. GH deficiency diagnosed by either of the following two criteria:

   1. . Peak GH response to L-arginine stimulation test < 1.4 microg/L; or
   2. . Plasma IGF-1 level 1 SD below the expected median for age and body weight.
7. Availability of caregiver to oversee administration of medications.
8. Reasonable expectation for completion of outcome measures
9. Residence inside the United States

Exclusion Criteria:

1. History of pre-existing neurologic disease (such as epilepsy, brain tumors, meningitis, cerebral palsy, encephalitis, brain abscesses, vascular malformations, cerebrovascular disease, Alzheimer's disease, multiple sclerosis, or HIV-encephalitis)
2. History of premorbid disabling condition that interfere with outcome assessments
3. Contraindication to rhGH therapy. (hypersensitivity to rhGH or any of the components of the supplied product, including metacresol, glycerin, or benzyl alcohol)
4. Penetrating traumatic brain injury
5. Diabetes mellitus.
6. Obesity (BMI > 30).
7. Active infection.
8. Active malignant disease.
9. Acute critical illness, heart failure, or acute respiratory failure
10. Previous hospitalization for TBI > 1 day
11. Membership in a vulnerable population (prisoner)
12. Pregnancy. Women of childbearing age will be given a pregnancy test during screening to exclude pregnancy.
13. Lactating females

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramon R. Diaz-Arrastia, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center; Randi Dubiel, MD, Study Director — Baylor Health Care System
Locations (3):
- United States (3):
  - Center for NeuroSkills, Bakersfield, California
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Treatment With Recombinant Human Growth Hormone: The GH treatment arm will receive a starting dose of 400 microgramsg/day, with increases (or decreases) in dose by 100-200 micrograms/day each month, monitoring for side effects, until goal IGF-1 (in the upper quartile of the range for age and body weight) is reached up to maximum dose of 1,000 microgramsg/day. Dose adjustments may be modified by the investigators for participants receiving oral estrogens or other circumstances know to influence GH dosing or atypical responses to treatment.
  Recombinant human Growth Hormone: 400 micrograms/day SC for 6 months. Dose adjusted based on serum IGF-1 measurements
- Placebo Treatment: Doses for participants receiving placebo will also be adjusted monthly to maintain the blinding.
  Placebo: SC injection daily
Period: Overall Study
Arm/Group | Active Treatment With Recombinant Human Growth Hormone | Placebo Treatment
Started | 31 | 32
Completed | 16 | 18
Not Completed | 15 | 14
Not completed — Lost to Follow-up | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Treatment With Recombinant Human Growth Hormone: The GH treatment arm will receive a starting dose of 400 microgramsg/day, with increases (or decreases) in dose by 100-200 micrograms/day each month, monitoring for side effects, until goal IGF-1 (in the upper quartile of the range for age and body weight) is reached up to maximum dose of 1,000 microgramsg/day. Dose adjustments may be modified by the investigators for participants receiving oral estrogens or other circumstances know to influence GH dosing or atypical responses to treatment.
  Recombinant human Growth Hormone: 400 micrograms/day SC for 6 months. Dose adjusted based on serum IGF-1 measurements
- Total: Total of all reporting groups
Arm/Group | Treatment With Recombinant Human Growth Hormone | Placebo Treatment | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (15.2) | 30.1 (13.7) | 31.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 28 | 30 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Dallas, Texas
  Participants
    United States | 31 | 32 | 63
Baseline IGF-1 level < 1 SD below expected mean [Count of Participants; unit: Participants] | 3 | 3 | 6
Baseline L-Arginine stimulation test [Median (Inter-Quartile Range); unit: ng/mL] | 2.2 [0.6 to 5.9] | 1.2 [0.5 to 5.7] | 1.3 [0.5 to 5.8]

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcome 6 Months After Injury, as Measured by the Processing Speed Index
Description: Processing Speed Index ages standardized score. In this scale, higher scores represent better functioning, lower scores represent poorer function.
  100 = mean of a normative population. 110 = 1 standard deviation above normal; 90 = 1 standard deviation below normal 120 = 2 standard deviations above normal; 80 = 2 standard deviations below normal
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Processing speed index standardized scor
Groups:
- rhGH Treatment: The GH treatment arm will receive a starting dose of 400 microgramsg/day, with increases (or decreases) in dose by 100-200 micrograms/day each month, monitoring for side effects, until goal IGF-1 (in the upper quartile of the range for age and body weight) is reached up to maximum dose of 1,000 microgramsg/day. Dose adjustments may be modified by the investigators for participants receiving oral estrogens or other circumstances know to influence GH dosing or atypical responses to treatment.
  Recombinant human Growth Hormone: 400 micrograms/day SC for 6 months. Dose adjusted based on serum IGF-1 measurements
- Placebo Treament: Doses for participants receiving placebo will also be adjusted monthly to maintain the blinding.
  Placebo: SC injection daily
Arm/Group | rhGH Treatment | Placebo Treament
Number analyzed (Participants) | 31 | 32
Processing speed index standardized scor | 82.5 [73.0 to 96.0] | 82.5 [79.0 to 99.0]

2. Secondary Outcome: IGF-1 Levels.
Description: Serum levels of Insulin-Like Growth Factor-1.
Time Frame: 4 years
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Active Treatment With Recombinant Human Growth Hormone | Placebo Treatment
Number analyzed (Participants) | 31 | 32
ng/mL | 245.5 [203.5 to 321.5] | 173.0 [145.0 to 237.0]

3. Secondary Outcome: Processing Speed Index 1 Year After Injury
Description: as for outcome 1
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: Processing speed index standardized scor
Arm/Group | Active Treatment With Recombinant Human Growth Hormone | Placebo Treatment
Number analyzed (Participants) | 31 | 32
Processing speed index standardized scor | 86.0 [76.0 to 111] | 89.5 [81.0 to 99]

4. Secondary Outcome: GH Response to L-arginine Stimulation at Baseline
Description: Measurement of serum GH levels over 90 minutes after administration of L-arginine
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Active Treatment With Recombinant Human Growth Hormone | Placebo Treatment
Number analyzed (Participants) | 31 | 32
ng/mL | 2.2 [0.6 to 5.9] | 1.2 [0.5 to 5.7]

5. Secondary Outcome: IGF-1 Levels
Description: Serum IGF-1 levels at baseline for both treatment groups was correlated with the Processing Speed Index recorded at baseline, using Pearson's correlation coefficient. Perason's correlation coefficient is a measure of the linear correlation between two variables X and Y. It has a value between +1 and -1, where 1 is total positive linear correlation, 0 is no linear correlation, and -1 is total negative linear correlation.
Time Frame: Baseline
Measure: Number; unit: Pearson's correlation coefficient
Arm/Group | Active Treatment With Recombinant Human Growth Hormone | Placebo Treatment
Number analyzed (Participants) | 31 | 32
Pearson's correlation coefficient | 0.1 | 0.1

6. Secondary Outcome: Rates of Diabetes Mellitus, Arthralgias, or Peripheral Edema.
Description: Rates of diabetes mellitus, arthralgias, or peripheral edema between rhGH treatment and placebo.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment With Recombinant Human Growth Hormone | Placebo Treatment
Number analyzed (Participants) | 31 | 32
Participants
  Diabetes mellitus | 0 | 0
  Arthralgia | 2 | 6
  Peripheral edema | 0 | 1
  None | 29 | 25

ADVERSE EVENTS:
Groups:
- Recombinant Human Growth Hormone: The GH treatment arm will receive a starting dose of 400 microgramsg/day, with increases (or decreases) in dose by 100-200 micrograms/day each month, monitoring for side effects, until goal IGF-1 (in the upper quartile of the range for age and body weight) is reached up to maximum dose of 1,000 microgramsg/day. Dose adjustments may be modified by the investigators for participants receiving oral estrogens or other circumstances know to influence GH dosing or atypical responses to treatment.
  Recombinant human Growth Hormone: 400 micrograms/day SC for 6 months. Dose adjusted based on serum IGF-1 measurements
Arm/Group | Recombinant Human Growth Hormone | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 2/31 | 2/32
Other Adverse Events (participants affected / at risk) | 12/31 | 15/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant Human Growth Hormone (N=31) | Placebo Treatment (N=32)
seizure (Nervous system disorders) | 2 | 2 — Patients with TBI are at high risk for post-traumatic seizures. Seizure in participants in this study are an expected adverse event
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Growth Hormone (N=31) | Placebo Treatment (N=32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Headache (Nervous system disorders) | 1 (31) | 3 (32)
Elective Surgery (General disorders) | 6 (31) | 4 (32)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (31) | 6 (32)
Drowsiness (Nervous system disorders) | 1 (31) | 1 (32)
Dry mouth (General disorders) | 1 (31) | 3 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No